CLINICAL TRIAL: NCT04999852
Title: The Effects of the Safe and Sound Protocol on PTSD Symptoms and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Spencer Psychology (Unknown)
Responsible Party: Principal Investigator, Jacek Kolacz, Research Fellow, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11261, 14850
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Post Traumatic Stress Disorder; Anxiety
Keywords: Post Traumatic Stress Disorder; Anxiety; PTSD treatment; Safe and Sound Protocol; SSP; auditory intervention; music intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Psychotherapy + SSP (Experimental): All subjects enrolled in this study will receive the SSP intervention
  Interventions: Device: Safe and Sound Protocol; Behavioral: Psychotherapy
- Psychotherapy (treatment as usual) (Active Comparator): Subjects who are receiving psychotherapy but not the SSP intervention
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Device: Safe and Sound Protocol — SSP is a non-invasive acoustic vagus nerve stimulator consisting of 5 hours of filtered and processed music designed to promote efficient regulation of autonomic state, and available through an app. The SSP is delivered via a mobile app and may fall under the heading of medical devices under the category of software functions/mobile medical applications.
  Other Names: SSP
  Arms: Psychotherapy + SSP
Behavioral: Psychotherapy — All participants, regardless of study arm, will be recruited from the pool of Spencer Psychology clients who are actively recieving psychotherapy. Participants will continue to recieve psychotherapy during the course of the study.

SUMMARY:
The Safe and Sound Protocol (SSP) is a passive acoustic intervention that is designed as a "neural exercise" to promote efficient regulation of autonomic state. Prior research has shown that the SSP can improve autonomic function, auditory hypersensitivities, and emotion regulation in individuals with Autism Spectrum Disorders. This observational pilot study is being conducted to establish methods for an upcoming randomized controlled trial to test the utility of the SSP for trauma treatment.

This study will enroll clients at the Spencer Psychology clinic who are set to take part in SSP under the supervision of their therapist. Because the therapists have participated in the design of the protocol and will participate in data collection and analysis, SSP will be considered a research procedure. In addition to taking part in SSP, subjects complete a set of questionnaires and have their pulse measured before starting the SSP intervention, after having completed 2/5 hours of the SSP, one week after completing all 5 hours of the SSP, and one month after completing the SSP intervention. The investigators will also pull relevant information from Spencer Psychology's medical records to document diagnosis, track client progress during study, and augment self-reported demographics. Clients who are receiving psychotherapy but not the SSP will be recruited as a comparison group.

ELIGIBILITY:
SSP Intervention Arm:

Inclusion Criteria:

* Client at Spencer Psychology in Bloomington, Indiana
* Diagnosed with PTSD or trauma not otherwise specified
* Already have agreed with therapist to administer SSP as a part of therapy

Exclusion Criteria:

* Tinnitus or hearing loss
* Diagnosed with cardiac arrhythmia
* At high risk for 2019 novel coronavirus (COVID-19) complications based on Center for Disease Control (CDC) guidelines, unless vaccinated

Comparison (Treatment As Usual) Arm Additional Criteria:

Inclusion Criteria:

1. 18 years of age or older
2. Active psychotherapy client at Spencer Psychology
3. Diagnosis of PTSD or trauma not otherwise specified
4. Match range of PCL-5 baseline scores with treatment arm during screener survey

Exclusion criteria:

1. Currently using or have previously used the Safe and Sound Protocol (SSP) in therapy
2. Current therapy includes Eye Movement Desensitization and Reprocessing (EMDR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kolacz, PhD, Principal Investigator — Indiana University
Locations (1):
- Spencer Psychology, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in using IPD collected or generated as part of this study may do so by contacting the study PI. Researchers will be asked to complete a Data Use Request Form, which includes contact information, description of the research project for which the data and/or code would be used, specification of which data and/or code would be needed for their proposed project, an approximate time line for their proposed project, and authorship on their proposed project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of primary results
Access Criteria: All requests for data will be reviewed by the PIs and co-Is and a majority vote will be used to determine whether the request is approved or not. If the request is approved, Dr. Kolacz will inform the requestor, return a signed copy of the completed Data Use Request Form to the requestor, and let the requestor know that written IRB approval of the requestor's proposed study from the requestor's home institution will be required before data and/or code will be shared with the requestor. If a request is approved pending revision to the Data Use Request Form, Dr. Kolacz will work with requestors to revise sections of their Data Use Request Forms in order to obtain approval. If the request is not approved, Dr. Kolacz will inform the requestor and returned a signed copy of the completed Data Use Request Form to the requestor that includes an explanation for the denial.

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychotherapy + SSP: All subjects enrolled in this study will receive the SSP intervention
  Safe and Sound Protocol: SSP is a non-invasive acoustic vagus nerve stimulator consisting of 5 hours of filtered and processed music designed to promote efficient regulation of autonomic state, and available through an app. The SSP is delivered via a mobile app and may fall under the heading of medical devices under the category of software functions/mobile medical applications.
  Psychotherapy: All participants, regardless of study arm, will be recruited from the pool of Spencer Psychology clients who are actively receiving psychotherapy. Participants will continue to receive psychotherapy during the course of the study.
- Psychotherapy (Treatment as Usual): Subjects who are receiving psychotherapy but not the SSP intervention
  Psychotherapy: All participants, regardless of study arm, will be recruited from the pool of Spencer Psychology clients who are actively receiving psychotherapy. Participants will continue to receive psychotherapy during the course of the study.
Period: Overall Study
Arm/Group | Psychotherapy + SSP | Psychotherapy (Treatment as Usual)
Started | 32 | 13
Completed | 19 | 12
Not Completed | 13 | 1
Not completed — Withdrawal by Subject | 11 | 1
Not completed — Switched to different psychotherapy that was ineligible for study | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Psychotherapy + SSP: Safe and Sound Protocol: SSP is a non-invasive acoustic vagus nerve stimulator consisting of 5 hours of filtered and processed music designed to promote efficient regulation of autonomic state, and available through an app. The SSP is delivered via a mobile app and may fall under the heading of medical devices under the category of software functions/mobile medical applications.
  Psychotherapy: All participants, regardless of study arm, will be recruited from the pool of Spencer Psychology clients who are actively receiving psychotherapy. Participants will continue to receive psychotherapy during the course of the study.
- Total: Total of all reporting groups
Arm/Group | Psychotherapy + SSP | Psychotherapy (Treatment as Usual) | Total
Number analyzed (Participants) | 32 | 13 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (13.7) | 36.2 (8.72) | 35.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 12 | 38
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 10 | 41
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post Traumatic Stress Disorder Symptoms
Description: Change in PTSD symptoms from baseline, measured using the Post Traumatic Stress Disorder Checklist for the DSM-5 (PCL-5), a 20-item self report. Total symptom severity scores range from 0 to 80, with higher scores indicating higher symptomology (poorer outcome).
Time Frame: 2-4 months. SSP Arm/Group assessed at baseline and 1 week after completion of the SSP intervention; Psychotherapy (Treatment as Usual) Arm/Group assessed at 3 months post-baseline (estimated average time to complete listening in SSP arm).
Population: Results are change scores from intent-to-treat analysis in which the last observed value is carried forward
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychotherapy + SSP | Psychotherapy (Treatment as Usual)
Number analyzed (Participants) | 32 | 13
score on a scale | -9.9 (11.1) | -2.3 (12.2)

2. Primary Outcome: Change From Baseline in Anxiety Symptoms
Description: Change from baseline in anxiety symptoms, measured using the Generalized Anxiety Disorder scale (GAD-7), 7-item self report. Scores range from 0-21 points, with higher scores indicating greater anxiety symptoms (poorer outcome).
Time Frame: as for outcome 1
Population: Intent to treat analysis with last observed value carried forward
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychotherapy + SSP | Psychotherapy (Treatment as Usual)
Number analyzed (Participants) | 32 | 13
score on a scale | -1.9 (3.5) | -0.8 (3.4)

3. Secondary Outcome: Change From Baseline in Self-reported Disruption of Autonomic Reactivity
Description: Change from baseline in autonomic symptoms, measured using the Body Perception Questionnaire (BPQ), 20-item self-report. T Scores (M = 50, SD = 10) were used, with higher scores indicating greater level of symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychotherapy + SSP | Psychotherapy (Treatment as Usual)
Number analyzed (Participants) | 32 | 13
score on a scale | -1.7 (5.5) | -0.1 (5.2)

4. Secondary Outcome: Change From Baseline in Mean Heart Period During Posture Shifts [SSP Arm Only]
Description: Change from baseline in mean heart period during supine, sitting, and standing posture shifts. Data was measured using an earlobe pulse sensor (Photoplethysmography). Longer heart period (higher values, reported in milliseconds) are indicative of lower autonomic arousal states. This metric is intended as a measure of mechanism and and high values may be associated with a better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Psychotherapy + SSP
Number analyzed (Participants) | 29
milliseconds
  Supine | -99.8 (117.0)
  Sitting | -90.0 (134.0)
  Standing | -70.2 (142.)

5. Secondary Outcome: Change From Baseline in Respiratory Sinus Arrhythmia (RSA) During Posture Shifts [SSP Arm Only]
Description: Change from baseline in Respiratory sinus arrhythmia (RSA) - a component of heart rate variability - measured during supine, sitting, and standing posture shifts. Measurements were conducted using an earlobe pulse sensor (Photoplethysmography). Greater RSA (higher values, reported in ln[milliseconds]^2) is associated with greater parasympathetic activity, which can help reduce physiological threat responses. This metric is intended to measure mechanism and high values may be associated with a better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln[milliseconds]^2
Arm/Group | Psychotherapy + SSP
Number analyzed (Participants) | 29
ln[milliseconds]^2
  Supine | -.35 (1.00)
  Sit | -.43 (1.44)
  Stand | -.04 (1.33)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked over the course of participation in the study (SSP+Psychotherapy Median Length = 145 days, Control Arm Median length = 122 days)
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Terms
Arm/Group | Psychotherapy + SSP | Psychotherapy (Treatment as Usual)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/13
Other Adverse Events (participants affected / at risk) | 1/32 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychotherapy + SSP (N=32) | Psychotherapy (Treatment as Usual) (N=13)
Other (Not Including Serious) Adverse Event (General disorders) | 1 (1) | 0 (0) — One participant felt increased anxiety and mild nausea following an SSP listening session. The client reported the event lasted about fifteen minutes, and then quickly dissipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT04999852/Prot_SAP_001.pdf